CLINICAL TRIAL: NCT03858725
Title: A Randomized, Open-label, Fasted, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-374 5 mg in Healthy Volunteer
Brief Title: Clinical Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-374 5 mg in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 190BE18031
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D569/CKD-374 5mg (Experimental): 1. Period 1: D569 Tab. 1T
  2. Period 2: CKD-374 5mg Tab. 1T
  Interventions: Drug: D569 Tab.; Drug: CKD-374 5mg Tab.
- CKD-374 5mg/D569 (Experimental): 1. Period 1: CKD-374 5mg Tab. 1T
  2. Period 2: D569 Tab. 1T
  Interventions: Drug: D569 Tab.; Drug: CKD-374 5mg Tab.

INTERVENTIONS:
Drug: D569 Tab. — D569 Tab. 1T single oral administration under fasting condition
Drug: CKD-374 5mg Tab. — CKD-374(Tofacitinib) 5mg Tab. 1T single oral administration under fasting condition

SUMMARY:
This study is a randomized, open-label, fasted, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-374 5 mg in healthy volunteers.

DETAILED DESCRIPTION:
To healthy subjects of thirty-six (36), following treatments are administered dosing in each period and wash-out period is a minimum of 7 days.

Reference drug: D569 Tab. / Test drug: CKD-374 5mg Tab. Pharmacokinetic blood samples are collected up to 12hrs. The pharmacokinetic characteristics and safety are assessed

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject older than 19 years and less than 55 years at the screening
2. Individuals who had 17.5 kg/m2 ≤ Body Mass Index(BMI) < 30.5kg/m2 and a total body weight ≥ 55 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Individuals who were deemed to be appropriate as study subjects in accordance with the screening results (laboratory tests, vital signs, ECG, chest X-ray etc.)
5. Individuals who signed an informed consent form approved by the IRB of Chonbuk National University Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content and characteristics of the investigational drug
6. Individuals with the ability and willingness to participate during the study period

Exclusion Criteria:

1. Individuals with a medical evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or immune disease (excluding simple dental history such as dental calculus, impacted tooth, wisdom tooth, etc.)
2. Individuals with a medical history of gastrointestinal disease (e.g., gullet disease including esophageal achalasia, esophagostenosis, or Crohn's disease) or operations (excluding simple appendectomy, herniotomy, or tooth extraction surgery) that may affect drug absorption
3. Individuals with the following laboratory test results: ALT or AST > 2x the upper limit of the normal range
4. A history of regular alcohol consumption exceeding 210 g/week within the 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
5. Individuals who smoked more than 20 cigarettes per day within 6 months prior to screening
6. Individuals who had been administered investigational product(s) of other clinical study or bioequivalence study within the 3 months prior to the first dose of this study
7. Individuals with the following vital signs results at screening

   *Individuals who had sitting blood pressure ≥90 mmHg or <140 mmHg (systolic) or ≥90 mmHg or <60 mmHg (diastolic)
8. Individuals with a medical history of significant alcohol abuse or drug abuse within one year prior to the screening
9. Individuals who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first dose of investigational product(s)
10. Individuals who had taken prescription or nonprescription drugs within the 10 days prior to the first dose of investigational product(s)
11. Individuals who donated whole blood within the 2 months, or blood components within 1 month prior to the first dose of the investigational product(s)
12. Individuals with severe acute/chronic medical or psychiatric conditions that may increase the risk associated with study participation or investigational product(s) administration, or may interfere with the interpretation of study results
13. Individuals with hypersensitivity to ingredients used in the investigational product(s)
14. Patients with serious infection (e.g., Sepsis) or active infection including localized infection or history of interstitial pneumonia
15. Patients with active tuberculosis or history of tuberculosis
16. Patients with hepatopathy
17. Patients with an absolute neutrophil count (ANC) less than 1000 /ul
18. Patients with an absolute lymphocyte count (ALC) less than 500 /ul
19. Patients who have hemoglobin levels less than 9 g/dL
20. Women who are pregnant or may be pregnant
21. Patients with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
22. Patients with nephropathy (eGFR<60 ml/min/1.73 m2)
23. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-374 and D569 | [Time Frame: Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours]
  Area under the CKD-374/ D569 concentration in blood-time curve from zero to final
Cmax of CKD-374 and D569 | [Time Frame: Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours]
  The maximum CKD-374/ D569 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Ho Jang, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No